CLINICAL TRIAL: NCT02047448
Title: Improving Medication Adherence Through a Transitional Care Pharmacy Practice Model
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wilkes University (Other)
Collaborators: Moses Taylor Hospital Foundation (Unknown); Commonwealth Health (Unknown); Community Pharmacy Foundation (Other)
Responsible Party: Principal Investigator, Judith L. Kristeller, Associate Professor, Wilkes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CPF
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Heart Failure
Keywords: transition of care; care transitions; readmission; medication; adherence; medication management; medication reconciliation; patient counseling; pharmacist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): The control group will receive the current standard of care including medication reconciliation during hospitalization performed by a nurse or physician and education about discharge medications provided by the inpatient nurse. There will not be a pharmacist discharge care plan developed for this group. The patients will not be required to choose a participating community pharmacist and no counseling and education appointments will be scheduled. Any medication-related problems identified by the pharmacists and will be communicated as appropriate and resolved as is the standard of care. Any other interaction between the patient and their pharmacist will be according to the current standard of care.
- Pharmacist Counseling (Experimental): The hospital pharmacist will meet with the patient and complete medication reconciliation, assess the patient's understanding of the medications, and identify medication-related problems. The hospital pharmacist will complete a pharmacist discharge care plan and a copy will be sent to the participating community pharmacist. The patients will be scheduled for the first meeting with their community pharmacist within 1 week of hospital discharge. The community pharmacist will interview the patient about their general health and any current symptoms of heart failure or COPD, identify any additional medication-related problems, follow-up on any issues as described in the pharmacist discharge care plan, and provide patient education. The patients will then meet with their community pharmacist for counseling and patient education at monthly intervals for 6 months following hospital discharge.
  Interventions: Procedure: Pharmacist Counseling

INTERVENTIONS:
Procedure: Pharmacist Counseling — The hospital pharmacist will meet with the patient and complete medication reconciliation, assess the patient's understanding of the medications, and identify medication-related problems. The hospital pharmacist will complete a pharmacist discharge care plan and a copy will be sent to the participating community pharmacist. The patients will be scheduled for the first meeting with their community pharmacist within 1 week of hospital discharge. The community pharmacist will interview the patient about their general health and any current symptoms of heart failure or COPD, identify any additional medication-related problems, follow-up on any issues as described in the pharmacist discharge care plan, and provide patient education. The patients will then meet with their community pharmacist for counseling and patient education at monthly intervals for 6 months following hospital discharge.
  Arms: Pharmacist Counseling

SUMMARY:
The purpose of this pilot study is to determine if medication adherence is improved by a transitional care pharmacy practice model designed to integrate hospital and community pharmacists in the care and education of patients with heart failure or COPD who are discharged from a community hospital to home. The hospital and community pharmacists will collaborate with each other, the patient, and other practitioners including the primary care physician, nurse, and case manager to prevent and correct medication-related problems and attempt to improve patient outcomes especially during the error-prone transition from hospital to home.

ELIGIBILITY:
Inclusion Criteria:

* admitted to hospital with a primary or secondary diagnosis of heart failure or COPD
* anticipated eventual discharge to home
* agreeable to participate in monthly counseling sessions (if randomized to intervention group) from a participating community pharmacist

Exclusion Criteria:

* presence of cognitive impairment or dementia that would significantly prevent effective patient education and counseling
* non English-speaking
* anticipated discharge to a long-term care or skilled nursing facility on a permanent basis
* permanent long-term care facility residents
* surgical patients
* hospice patients
* patients who die within 30 days of initial study hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-01; Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Medication Adherence | 6 months
  The primary endpoint will be medication adherence as measured by the Proportion of Days Covered (PDC) calculation. This is calculated by dividing the total days' supply dispensed by 180 days. Medications considered in this calculation will include those used for the treatment of heart failure or COPD and known to improve outcomes. The composite PDC will be an average of the individual PDC for each drug class.

SECONDARY OUTCOMES:
Medication related problems | 6 months
  Actual or potential medication-related problems (MRP) that are identified by the hospital and participating community pharmacists will be categorized based on an MRP classification tool.
Patient Satisfaction | 6 months
  The Care Transitions Measure (CTM-3) is a validated survey to assess the patient's satisfaction with the quality of transitional care during hospitalization and will be completed by the patient following hospital discharge. The patient's satisfaction with the services provided by the community pharmacies will be assessed with the Consumer Experience with Pharmacy Services survey (© Pharmacy Quality Alliance).
Hospital readmissions or ED visits | 6 months
  Hospital readmissions are defined as an unplanned and overnight admission to the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Judith Kristeller, PharmD, Principal Investigator — Wilkes University
Locations (1):
- Moses Taylor Hospital, Scranton, Pennsylvania, United States